CLINICAL TRIAL: NCT07061548
Title: Development of an Artificial Intelligence Model for Predicting Intraoperative Changes in Cardiac Output Using Capnography During General Anesthesia
Brief Title: Algorithm Predicting Intraoperative Changes in Cardiac Output Using Capnography
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Heejoon Jeong, Clinical Assistant Professor, Samsung Medical Center
Other Study IDs: SMC2025-06-120-001
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: General Anesthesia Using Endotracheal Intubation
Keywords: artificial intelligence; general anesthesia; capnography; cardiac output

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- capnography-cardiac output cohort: Adult patients who underwent surgery under general anesthesia with capnography and invasive arterial blood pressure monitor
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No intervention

SUMMARY:
Conventional monitoring of cardiac output requires an invasive procedure and an additional device, which can lead to increased risk and cost. Investigators developed an artificial intelligence algorithm to predict intraoperative changes in cardiac output using capnography in patients undergoing surgery under general anesthesia.

DETAILED DESCRIPTION:
Anesthesiologists strive to maintain adequate cardiac output during surgery. However, conventional monitoring of cardiac output requires an invasive procedure (risk) and an additional device (cost).

Because most surgeries are performed without any invasive monitors, anesthesiologists must manage the patients without cardiac output information.

However, modern anesthesia machines usually provide capnography, and continuous capnography monitoring can help estimate changes in cardiac output. Therefore, investigators aim to develop an artificial intelligence algorithm to predict intraoperative changes in cardiac output using capnography in patients undergoing surgery under general anesthesia.

Investigators train a model using capnography data (5-minute duration) related to a 20% or greater decrease in cardiac output during the same period. The developed model can provide an alarm for a decrease in cardiac output based on the change in capnography.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery under general anesthesia
* Adult patients (18 < age < 76)
* Patients who were monitored invasive arterial blood pressure (waveform) and capnography (numeric)

Exclusion Criteria:

* Emergency surgery
* Cardiovascular and thoracic surgery
* Known Asthma and Chronic obstructive pulmonary disease (COPD)
* Preoperative pulmonary function test (PFT) abnormality over moderate grade
* Intraoperative monitoring duration less than 30 minutes

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient who underwent surgery under general anesthesia in Samsung Medical Center, Seoul, South Korea
Sampling Method: Non-Probability Sample
Enrollment: 2005 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Predictability of algorithm | Every time points with interval of 5 minutes during surgery
  The performance of the algorithm to predict whether cardiac output has decreased by more than 20% compared to 5 minutes ago. Predictability is estimated by area under the receiver-operating characteristic curve analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided